CLINICAL TRIAL: NCT03717480
Title: A Phase 2 Study of Ex Vivo TCR αβ T Cell Depletion for Graft-Versus-Host Disease (GVHD) Prophylaxis in Mismatched Donor Peripheral Blood Stem Cell Transplantation for Hematologic Malignancies
Brief Title: Ex Vivo TCR αβ T Cell Depletion for Graft-Versus-Host Disease Prophylaxis in Mismatched Donor Peripheral Blood Stem Cell Transplantation for Hematologic Malignancies
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was prematurely closed to enrollment due to feasibility issues, as the site has promising upcoming competing trials, and the study was already not enrolling at a rate sufficient to meet the accrual goal.
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Vincent T. Ho, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-270
Record Dates: First submitted 2018-10-22; First posted 2018-10-24 (Actual); Results first posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-04

CONDITIONS: Hematologic Malignancy
Keywords: Graft vs. Host Disease; Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms; Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- TCR α/β Reagent System (Experimental): * The stem cell apheresis product will be depleted of TCRαβ T cells by negative selection using the automated CliniMACS® Plus device.
  * CD34+ stem cell counts will be obtained before and after processing with the Miltenyi ClinicMACs device
  Interventions: Device: ClinicMACs

INTERVENTIONS:
Device: ClinicMACs — The Reagent System will remove certain cells (called T-Cell Receptor (TCR) α/β positive T-cells) that are thought to cause GVHD from donor product before it is given to participants

SUMMARY:
This research study is studying the removal of a subset of white blood cells (called alpha/beta T cells) from the donor product using a cell separation device before the product is transplanted into the participant.

The device used to remove the α/βT cells in this study is:

-CliniMACS® TCR α/β Reagent System

DETAILED DESCRIPTION:
Patients who receive an allogeneic (using another person as the donor) stem cell transplant (SCT) are at risk for developing graft-versus-host disease (GVHD).

The word "graft" refers to the donor blood cells that you will receive during the transplant. The word "host" refers to the person receiving the cells. GVHD is a complication of transplantation where the donor graft attacks and damages some of the participant's tissues.

GVHD may occur when the T cells (a type of white blood cell that helps protect the body from infection) from the donor react against normal tissues or organs in the body. There are two basic types of GVHD:

* Acute GVHD often occurs early (generally first 3-6 months after SCT) may affect skin, gastrointestinal tract (stomach and intestines) and liver.
* Chronic GVHD often occurs later (Usually after 3-6 months after SCT) and may affect many organs and significantly diminish quality of life.

To confirm the diagnosis of acute or chronic GVHD, the participant may be asked to have a biopsy (a small sample of the participant's tissue to look at under the microscope) of the skin, gut, or, rarely, the liver.

In this research study, the investigator are investigating a pre-transplant intervention aimed to prevent GVHD by processing the donor product with the Miltenyi CliniMACS TCR α/β Reagent System. The Reagent System will remove certain cells (called T-Cell Receptor (TCR) α/β positive T-cells) that are thought to cause GVHD from donor product before it is given to the participant. By selectively removing this specific type of T cells from the donor product, the investigators hope to reduce the risk for GVHD without reducing the efficacy of the transplant.

This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved CliniMACS α/β T cell depletion system for use in the US, but this system is approved by the European Medicines Agency (EMA) and used in Europe

ELIGIBILITY:
Inclusion Criteria:

* Diagnoses and stage at time of transplant admission:

  * Acute leukemia (AML or ALL or MPAL) in first or subsequent remission
  * Myelodysplastic syndromes (MDS) with <10% marrow blasts
  * Myeloproliferative neoplasm (MPN) with <10% marrow blasts
  * CMML with less than 10% marrow blast
  * CML accelerated phase or second or subsequent chronic phase
  * Non-Hodgkin's lymphoma in PR or CR2 or beyond
  * Hodgkin lymphoma in PR or CR2 or beyond
* Age 18-65 years
* Patient has a related or unrelated donor who is 8 or 9 out of 10 match at HLA A, B, C, DRB1 and DQB1, based on allele level typing.
* Patient ECOG performance status 0-2 (Karnofsky ≥60%, see Appendix A)
* Patient deemed to be appropriate candidate for myeloablative conditioning transplantation.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patient with active HIV infection
* Chronic active hepatitis B infection (HepB surface Ag+ or detectable Hep B viral load)
* Prior allogeneic hematopoietic stem cell transplantation
* Impaired cardiac function- ejection fraction < 40%
* Impaired pulmonary function- pretransplant FEV1, DLCO < 50%
* Impaired renal function, based on

  --Serum creatinine > 2.0 mg/dl
* Impaired liver function unrelated to primary disease, based on

  --ALT or AST > 3x ULN, or Total Bilirubin > 2.0mg/dl (with exception for known or suspected Gilbert's disease)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Women who are pregnant or breast feeding. Women of child bearing potential must have a negative serum pregnancy test at study entry.
* Participants who are receiving any other investigational agents are eligible but such agent must be discontinued before admission for HSCT, and if resumption of investigation agent is planned after HSCT, this must be approved by the study PI.
* Participants with known active CNS disease. CNS disease that has been treated is eligible

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent T Ho, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- TCR α/β Reagent System: The stem cell apheresis product was depleted of TCRαβ T cells by negative selection using the automated CliniMACS® Plus device.
  CD34+ stem cell counts were obtained before and after processing with the Miltenyi ClinicMACs device.
  ClinicMACs: The Reagent System removed certain cells (called T-Cell Receptor (TCR) α/β positive T-cells) that are thought to cause GVHD from donor product before it was given to participants.
Period: Overall Study
Arm/Group | TCR α/β Reagent System
Started (Assignment to study arm) | 2
Receipt of Investigational Product/Study Treatment | 1
Completed (Survival to day 100 for evaluation of primary endpoint (severe acute GVHD-free survival rate)) | 1
Not Completed | 1
Not completed — Never received investigational product due to product viability limitations. | 1

BASELINE CHARACTERISTICS:
Population: Only evaluable participants, defined as participants who received investigational product, are included in the analysis population. Therefore, participants who never started protocol treatment have been excluded.
Arm/Group | TCR α/β Reagent System
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Severe Acute GVHD-free Survival
Description: Number of participants with severe acute GVHD-free survival will be assessed at 100 days post-SCT
Time Frame: 100 Days
Measure: Count of Participants; unit: Participants
Arm/Group | TCR α/β Reagent System
Number analyzed (Participants) | 1
Participants | 1

2. Secondary Outcome: Number of Participants With Grades II-IV Acute GVHD
Description: Grades II-IV acute GVHD will be assessed at 2 years post-SCT. Grade I GVHD is characterized as mild disease, grade II as moderate, grade III as severe, and grade IV as life-threatening. Higher grades of acute GVHD are associated with worse outcomes. Acute GVHD will be staged by assessment of clinical manifestations in the skin, gastrointestinal tract, and liver.
Time Frame: 2 years
Population: No participants were analyzed for this secondary outcome measure, because the only participant who would have been evaluable for analysis did not survive to the analysis timepoint of 2 years post-transplant.
Arm/Group | TCR α/β Reagent System
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants With Chronic GVHD
Description: Number of participants with chronic GVHD will be assessed at 2 years post-SCT.
Time Frame: 2 years
Population: as for outcome 2
Arm/Group | TCR α/β Reagent System
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants With GVHD and Relapse Free Survival (GRFS)
Description: GRFS will be defined as alive without having experienced grade III-IV acute GVHD, moderate/severe chronic GVHD, or relapse of underlying malignancy.
Time Frame: 2 years
Population: as for outcome 2
Arm/Group | TCR α/β Reagent System
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants With Immunosuppression-free Survival
Description: Number of participants with immunosuppression-free survival will be assessed at 2 years post-SCT.
Time Frame: 2 years
Population: as for outcome 2
Arm/Group | TCR α/β Reagent System
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Participants With Hematologic Recovery
Description: Hematologic recovery will be assessed in participants at 2 years post-SCT.
Time Frame: 2 years
Population: as for outcome 2
Arm/Group | TCR α/β Reagent System
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Participants With Immune Reconstitution
Description: Immune reconstitution will be assessed in participants at 2 years post-SCT.
Time Frame: 2 years
Population: as for outcome 2
Arm/Group | TCR α/β Reagent System
Number analyzed (Participants) | 0

8. Secondary Outcome: Number of Participants With Disease Relapse
Description: Disease relapse will be assessed in participants at 2 years post-SCT.
Time Frame: 2 years
Population: as for outcome 2
Arm/Group | TCR α/β Reagent System
Number analyzed (Participants) | 0

9. Secondary Outcome: Number of Participants With Transplant-related Mortality
Description: Participant transplant-related mortality will be assessed at 2 years post-SCT.
Time Frame: 2 years
Population: as for outcome 2
Arm/Group | TCR α/β Reagent System
Number analyzed (Participants) | 0

10. Secondary Outcome: Number of Participants With Organ Toxicity
Description: Participant organ toxicity will be assessed at 2 years post-SCT.
Time Frame: 2 years
Population: as for outcome 2
Arm/Group | TCR α/β Reagent System
Number analyzed (Participants) | 0

11. Secondary Outcome: Rates of Infections
Description: Participant rate of infections will be assessed at 2 years post-SCT.
Time Frame: 2 years
Population: as for outcome 2
Arm/Group | TCR α/β Reagent System
Number analyzed (Participants) | 0

12. Secondary Outcome: Number of Participants With Relapse-free and Overall Survival
Description: Number of participants with relapse-free and overall survival will be assessed at 2 years post-SCT.
Time Frame: 2 years
Population: as for outcome 2
Arm/Group | TCR α/β Reagent System
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for each participant up until 2 years post-transplant or until the participant's death, whichever came first. The only participant who received study treatment did not survive to the analysis timepoint of 2 years post-transplant, so all documented adverse events were collected from the date of their transplant up until their death approximately 9 months post-transplant.
Description: Adverse events were collected through regular investigator assessment and laboratory testing.
Arm/Group | TCR α/β Reagent System
All-Cause Mortality (participants affected / at risk) | 1/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TCR α/β Reagent System (N=1)
Hepatic Hemorrhage (Hepatobiliary disorders) | 1
Colonic Perforation (Gastrointestinal disorders) | 1
Platelet Count Decreased (Investigations) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Acute Kidney Injury (Renal and urinary disorders) | 1
Stroke (Nervous system disorders) | 1
Colitis (Gastrointestinal disorders) | 1 — Adenovirus
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TCR α/β Reagent System (N=1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 1 (3)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (2)
Aspartate Aminotransferase Increased (Investigations) | 1 (3)
Bacteremia (Infections and infestations) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Creatinine Increased (Investigations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (2)
Dizziness (Nervous system disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Infections and Infestations - Other, specify (Infections and infestations) | 1 (1) — EBV+
Mucositis Oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (3)
Platelet Count Decreased (Investigations) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2)
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Vaginal Pain (Reproductive system and breast disorders) | 1 (1)
Weight Loss (Investigations) | 1 (1)
White Blood Cell Decreased (Investigations) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination after accrual of only one evaluable subject resulted in an insufficient sample size for analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-08): https://cdn.clinicaltrials.gov/large-docs/80/NCT03717480/Prot_SAP_000.pdf